CLINICAL TRIAL: NCT06307314
Title: A Prospective Cohort Study of Plasma SAA1 Levels in Predicting Response to Radiotherapy-induced Oral Mucositis
Brief Title: Plasma SAA1 Levels in Predicting Response to Radiotherapy-induced Oral Mucositis
Status: Recruiting | Type: Observational
Sponsor: Nanfang Hospital, Southern Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: NFEC-2024-093
Record Dates: First submitted 2024-03-06; First posted 2024-03-12 (Actual); Last update posted 2024-03-12 (Actual); Status verified 2024-03

CONDITIONS: Nasopharyngeal Carcinoma; Head and Neck Cancer; Radiotherapy-induced Oral Mucositis; Biomarker
Keywords: SAA1; Radiotherapy-induced Oral Mucositis; Head and Neck Cancer; Nasopharyngeal Carcinoma
MeSH Terms: conditions — Nasopharyngeal Carcinoma; Head and Neck Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Tissue and plasma
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Head and neck squamous cell carcinoma (SCC) is the sixth most common cancer worldwide, with more than 700,000 new cases and more than 350,000 deaths each year. At present, radiotherapy is an important measure to control the recurrence of head and neck tumors, but almost all patients with head and neck squamous cell carcinoma will have acute inflammatory reactions such as radiotherapy-induced oral mucositis (RIOM) after radiotherapy, which seriously affects the quality of life and radiotherapy efficacy of patients. Serum amyloid A1 (SAA1) is an acute phase protein associated with inflammation. Our previous basic research found that serum SAA1 expression levels can be used as biomarkers to assess the dose received by the receptor in the early stages of radiation damage. At the same time, we confirmed that the serum level of SAA1 in patients with nasopharyngeal carcinoma increased after radiotherapy. Therefore, we intend to conduct a prospective, multicenter, observational study to further explore the predictive power of plasma SAA1 levels for radiotherapy-induced oral mucositis, with a view to early screening and prevention of RIOM patients.

ELIGIBILITY:
Inclusion Criteria:

* Over 18 years of age.
* Voluntarily sign informed consent.
* The pathological diagnosis was nasopharyngeal carcinoma, head and neck tumor.
* Need to be treated with radiotherapy.
* ECOG PS Score: 0/1.

Exclusion Criteria:

* There are contraindications to radiotherapy.
* Combined with other tumors.
* Patients had any serious coexisting medical conditions that could pose an unacceptable risk or negatively affect trial adherence. For example, unstable heart disease requiring treatment, chronic hepatitis, kidney disease, poor disease status, uncontrolled diabetes (fasting blood glucose > 1.5 × ULN), and mental illness.
* At the investigator's discretion, those who was not considered to be suitable for participation in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with nasopharyngeal carcinoma and head and neck tumors requiring radiotherapy.
Sampling Method: Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2024-02-01 (Actual); Primary Completion 2026-12-01 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Different grades radiotherapy-induced oral mucositis | Through study completion, up to 3 years
  The incidence different grades of radiotherapy-induced oral mucositis will be calculated.

SECONDARY OUTCOMES:
Start and duration of radiotherapy-induced oral mucositis | Through study completion, up to 3 years
  Calculated the onset time and duration of radiotherapy-induced oral mucositis.
Side effects of radiotherapy | Through study completion, up to 3 years
  Record other early or late side effects caused by radiotherapy.
Tumor response | Through study completion, up to 3 years
  The efficacy of tumor therapy was evaluated based on RECIST 1.1.

CONTACTS AND LOCATIONS:
Overall Officials: Jian Guan, Ph.D., Principal Investigator — Nanfang Hospital, Southern Medical University
Locations (5):
- China (5):
  - Nanfang hospital, Southern medical university, Guangzhou, Guangdong
  - Fujian Provinical Hospital, Fuzhou
  - Huizhou Central People's Hospital, Huizhou
  - Jieyang People's Hospital, Jieyang
  - Meizhou People's Hospital, Meizhou Academy of Medical Sciences Meizhou, Meizhou

IPD SHARING:
Plan to Share IPD: No